CLINICAL TRIAL: NCT06126419
Title: Application of High-Dose Insulin Therapy Using a Hyperinsulinemic Normoglycemic Clamp to Improve Liver Function and Regeneration
Brief Title: Application of High-dose Insulin Therapy to Improve Liver Function and Regeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, peter metrakos, Professor of Surgery, Program Leader - MUHC-RI Cancer Research Program, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-8880
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Liver Dysfunction; Liver Metastasis Colon Cancer; Liver Regeneration
Keywords: Hyperinsulinemic-Normoglycemic Clamp; High Dose Insulin Therapy; 99mTc-Mebrofenin Hepatobiliary Scintigraphy; Colorectal Cancer Liver Metastasis; Liver Resection
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: Group 1 will consist of participants scheduled for liver resection and will undergo high-dose insulin therapy preoperatively to determine if baseline liver function can be optimized/improved, as measured by 99mTc-Mebrofenin HBS. Cytokine profiling will also be collected and analyzed pre- and post-insulin infusion.
  Group 2 will consist of participants scheduled for liver resection that require LVD. They will then be randomized to two different arms -- control vs high-dose insulin therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Effect of high-dose insulin therapy on pre-operative liver function (Experimental): Group 1 will consist of participants scheduled for liver resection and will undergo high-dose insulin pre-operatively to determine if baseline liver function can be optimized/improved, as measured by 99mTc-Mebrofenin HBS.
  Interventions: Drug: High-Dose Insulin Therapy
- Group 2: Effect of high-dose insulin therapy on pre-operative liver function after LVD (Experimental): Group 2 will consist of participants scheduled for liver resection that require LVD. The participants in the experimental arm will receive high-dose insulin therapy after LVD.
  Interventions: Drug: High-Dose Insulin Therapy
- Group 3: Effect of high-dose insulin therapy on pre-operative liver function after LVD (No Intervention): Group 3 will consist of participants scheduled for liver resection that require LVD. The participants in the no intervention arm will not undergo intervention with high-dose insulin therapy after LVD.

INTERVENTIONS:
Drug: High-Dose Insulin Therapy — A baseline blood glucose value will be obtained. Two units of insulin will be administered IV if the blood glucose is > mmol/L. An insulin infusion of 0.12 units/kg/hr will be started. Ten minutes after starting the insulin, and when the blood glucose is < 6 mmol/L, dextrose 20% supplemented with phosphate (30 mmol/L) will be infused. Blood glucose levels will be measured every 15 minutes, and the dextrose infusion rate adjusted to maintain glycemic levels between 4 and 6 mmol/L for a duration of 6 hours. At the end of the 6 hour period, the insulin will be stopped and the dextrose will be weaned off.
  Arms: Group 1: Effect of high-dose insulin therapy on pre-operative liver function; Group 2: Effect of high-dose insulin therapy on pre-operative liver function after LVD

SUMMARY:
The primary objective of this interventional study is determine if the future liver remnant can be optimized by improving liver function pre-operatively in patients who are scheduled for major hepatectomy. The main questions it aims to answer are:

1. Does high-dose insulin therapy improve liver function in the pre-operative setting?
2. What is the effect of high-dose insulin therapy on liver function and liver regeneration after a liver venous deprivation (LVD) procedure?
3. What is the relationship between volume hypertrophy and function in the regenerating liver? Participants will receive a 6-hour infusion of insulin and dextrose to maintain a hyperinsulinemic-normoglycemic state in the weeks prior to planned liver surgery to assess its effect on liver function measured by 99m-Tc-Mebrofenin hepatobiliary scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Candidate for major liver resection
* Resectable colorectal liver metastasis

Exclusion Criteria:

* Inability to give consent
* Type 1 diabetes mellitus
* Uncontrolled blood glucose levels (fasting level > 10 mmol/L)
* Unresectable colorectal liver metastasis
* Extrahepatic metastatic disease that is unresectable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Liver function improvement after high-dose insulin therapy measured with 99mTc-Mebrofenin Hepatobiliary Scintigraphy (HBS). | Baseline to 24-hours post treatment
  99mTc-Mebrofenin HBS is a diagnostic nuclear medicine imaging procedure used to evaluate liver function by measuring radiotracer uptake and excretion. The outcome will be evaluating a measurable increase in 99mTc-Mebrofenin (measured %/min/meter^2) from baseline scan to post-treatment scan.
Liver function improvement after high-dose insulin therapy after LVD measured with 99mTc-Mebrofenin Hepatobiliary Scintigraphy (HBS). | Baseline to 7 days post treatment
  99mTc-Mebrofenin HBS is a diagnostic nuclear medicine imaging procedure used to evaluate liver function by measuring radiotracer uptake and excretion. The outcome will be evaluating a measurable increase in 99mTc-Mebrofenin (measured %/min/meter^2) from baseline scan to post-treatment scan.
Liver regeneration improvement after high-dose insulin therapy after LVD measured CT volumetry | Baseline to 7 days post treatment
  The volume of the liver can be measured from liver protocoled CT scans

CONTACTS AND LOCATIONS:
Locations (1):
- McGill Univeristy Health Centre, Montreal, Quebec, Canada